CLINICAL TRIAL: NCT05978336
Title: SuPA Mobility: Supporting Physical Activity for Mobility in Mobility-Limited Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H21-00858
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Limitation, Mobility; Older Adults
Keywords: physical activity; health coaching; exercise; limited mobility
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching (HC) (Experimental): The health coaching program will be delivered by trained and certified kinesiologists utilizing Brief Action Planning (BAP) principals. The BAP behavior change approach utilizes the following 4 techniques: 1) goal-setting; 2 )action planning; 3) self-monitoring; and 4) feedback. Participants will utilize daily physical activity diaries to enable self-monitoring, and BAP coaches will provide feedback on progress toward individualized physical activity goals.
  Interventions: Behavioral: Health Coaching Program
- Health Education Program (ED) (Active Comparator): This program is an attention control group, which consists of general health education. Education sessions will be delivered either by zoom or in person. The education sessions will cover the following topics: 1) falls prevention; 2) sleep; 3) healthy eating; 4) cognitive health; and 5) mental and emotional health.
  Interventions: Behavioral: Health Education Program

INTERVENTIONS:
Behavioral: Health Coaching Program — The HC program will be delivered over 26-weeks. Participants will have an initial hour-long HC session where the BAP coach will conduct a brief physical assessment and work with the participant to establish their physical activity goals and develop a plan. After the initial consult, coaches will conduct 8 x 20-minute phone calls with participants over the 26-week trial decreasing from bi-weekly phone calls in weeks 1-12 to monthly phone calls in weeks 13-26.
  Participants in the HC group will have an overall goal of increasing their weekly participation in moderate to vigorous physical activity by 50 minutes, via 5-, 7-, or 10-minute bouts of progressive exercises, at a rate of perceived exertion range of 13-14 ("somewhat hard") by week 16. Participants will have access to specific exercise sessions made available by YouTube and/or hardcopy manuals created by the research team.
  Other Names: HC
  Arms: Health Coaching (HC)
Behavioral: Health Education Program — Participants will begin with a one-hour, group-based, interactive education session on falls prevention delivered either in-person or by Zoom. Following the initial education session, ED participants will receive additional group education sessions (in-person or by Zoom) with the same duration and schedule as the HC program covering a variety of healthy aging topics.
  Other Names: ED
  Arms: Health Education Program (ED)

SUMMARY:
The goal of this randomized controlled trial is to investigate the effectiveness of a health-coaching intervention to improve physical activity in older adults with limited mobility when compared to a control, health education group.

DETAILED DESCRIPTION:
A total of 290 older adults with limited mobility will be randomized to either a 26-week health coaching program or health education program. Outcomes will be assessed at baseline, 13-weeks, 26-weeks (end of intervention), and 52 week (6-month follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* scored ≤ 9/12 on the SPPB
* are able to complete the 400-m walk in ≤ 15 minutes without sitting or physical assistance from another person or walker (use of cane is acceptable)
* scored 22/30 or higher on the Mini-Mental State Examination (MMSE)
* have no significant functional impairment as indicated by a score of 6/8 or higher on the Lawton and Brody Instrumental Activities of Daily Living Scale
* are able to safely engage in MVPA as indicated by the PAR-Q+ and by the family or study physician as necessary
* are community-dwelling
* are able to provide written informed consent.

Exclusion Criteria:

* are diagnosed with dementia or stroke
* self-report engaging in MVPA ≥ 10 minutes per week in the prior 3 months
* are unable to understand, speak, and read English proficiently

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mobility | Baseline, 13-weeks, 26-weeks, 52-weeks
  Measured by the Short Physical Performance Battery (SPPB)

SECONDARY OUTCOMES:
Physical activity | Baseline, 13-weeks, 26-weeks, 52-weeks
  Time spent moderate to vigorous physical activity and sedentary time measured by accelerometer.
Self reported physical activity | Baseline, 13-weeks, 26-weeks, 52-weeks
  Measured by the Community Health Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire for Older Adults.
Gait speed | Baseline, 13- weeks, 26-weeks, 52-weeks
  Measured during the 4-m walk
Capacity to complete the 400-m walk in ≤ 15 minutes | Baseline, 13- weeks, 26-weeks, 52-weeks
  measured as yes or no
Cognitive function | Baseline, 26-weeks, 52-weeks
  Measured with the NIH Toolbox and standard neuropsychological assessments
Community mobility | Baseline, 13-weeks, 26-weeks, 39-weeks, 52-weeks
  Measured with the Life Space Questionnaire
Functional mobility | Baseline, 13-weeks, 26-weeks, 39-weeks, 52-weeks
  Measured as the time to complete the Timed Up-and-Go (TUG)
Fatigue | Baseline, 13-weeks, 26-weeks, 39-weeks, 52-weeks
  Measured by the 9-item Fatigue Severity Scale (FSS) scored from 9 to 63, with higher scores indicating more severe fatigue
Lower extremity strength | Baseline, 13- weeks, 26-weeks, 52-weeks
  Measured with strain gauge (kilograms) on dominant quadriceps
Grip strength | Baseline, 13-weeks, 26-weeks, 52-weeks
  Measured with digital Jamar isometric dynamometer (Newtons)
Mood | Baseline, 13-weeks, 26-weeks, 39-weeks, 52-weeks
  Measured by the Centre for Epidemiological Studies Depression Scale (CES-D)
Health-related quality of life | Baseline, 13-weeks, 26-weeks, 39-weeks, 52-weeks
  Measured with questionnaire EuroQol (EQ-5D-5L)
Sleep | Baseline, 13-weeks, 26-weeks, 39-weeks, 52-weeks
  Measured with 19-item Pittsburgh Sleep Quality Index
Sleep | Baseline, 13-weeks, 26-weeks, 52-weeks
  Measured by accelerometer
Falls | Baseline, monthly
  Assessed with monthly calendar and questionnaire
Health resource utilization | Baseline, 13-weeks, 26-weeks, 39-weeks, 52-weeks
  Assessed with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health Research Institute Research Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rice J, Li LC, Davis JC, Pahor M, Madden K, Wei N, Wong H, Skelton DA, McCormick S, Falck RS, Barha CK, Rhodes RE, Loomba S, Sadatsafavi M, Liu-Ambrose T. Supporting physical activity for mobility in older adults with mobility limitations (SuPA Mobility): study protocol for a randomized controlled trial. Trials. 2023 Nov 28;24(1):769. doi: 10.1186/s13063-023-07798-9. PMID 38017467